CLINICAL TRIAL: NCT01496014
Title: Assessment of Severe Extremity Wound Bioburden at the Time of Definitive Wound Closure or Coverage: Correlation With Subsequent Post-Closure Deep Wound Infection: Bioburden Study
Brief Title: Assessment of Severe Extremity Wound Bioburden at the Time of Definitive Wound Closure or Coverage
Acronym: Bioburden
Status: Completed | Type: Observational
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: A-15737.5a
Record Dates: First submitted 2011-11-07; First posted 2011-12-21 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Open Fracture
Keywords: open fracture wounds; infections; tibia fractures; antibiotic therapies in severe fractures; All severe open fracture of the tibia bone
MeSH Terms: conditions — Fractures, Open; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- severe open fractures of the tibia bone

SUMMARY:
The purpose of this study is to characterize the bacteria in the wound "bioburden" at the time of definitive wound coverage/closure of severe tibia fractures in both the military and civilian populations.

DETAILED DESCRIPTION:
Infection remains the most common and significant complication following high energy fractures. The strategies used in the prevention of deep infection following severe open fracture wounds have remained constant for the past 20 years.

This project is designed to analyze the microbiology profiles of wounds from severe tibia fractures at closure by comparing two methods: routine microbiology techniques and PCR methods using the Ibis T5000 Biosensor System. The results from both identification methods will be compared to the pathogens associated with deep surgical site infections that occur post closure of the wound. Currently it is unknown which of these methods will yield information that can lower complication rates and better function of the leg. Our goal is to perform a multi-center, prospective cohort study of wound bacterial bioburden and associated antibiotic care in severe open lower extremity fractures.

Primary Aim: In a subset of 60 patients, compare the bioburden, as detected by Ibis technology, from each of three sampling techniques (deep tissue; soft tissue composite; composite of tissue from the length and depth of the wound). Samples obtained using the most effective technique identified in this step will be processed using Ibis in subsequent tissue analysis. Effectiveness is defined as the ability to identify key wound infection-causing pathogens.

Primary Hypothesis: The composite sampling approach will be the most effective technique.

Secondary Aim: Characterize the wound bioburden at the time of definitive wound closure or coverage using the Ibis T5000 Biosensor System PCR technology as compared to standard microbiology techniques.

Hypothesis 2: The Ibis technology will detect more species of pathogens than standard microbiology techniques. The percent of patients for whom Ibis will detect all species identified by standard microbiology will be greater than 95%.

Specific Aim 3: Characterize the wound bioburden in the patients who develop deep infection within one year of wound closure, and determine the association between infecting pathogens with initial wound closure bioburden as measured jointly by Ibis and standard microbiology techniques.

Specific Aim 4: Document the variability in antibiotic selection and duration, and examine the impact of this selection on subsequent deep infection.

Hypothesis 4a: Among patients treated with antibiotic regimens that are appropriate for the pathogens identified by standard microbiology, there will be a lower probability of deep infection than among those patients who received inappropriate antibiotic regimens.

Hypothesis 4b: Among patients treated with antibiotic regimens that are appropriate for the pathogens identified by Ibis, there will be a lower probability of deep infection than among those patients who received inappropriate antibiotic regimens.

ELIGIBILITY:
Inclusion Criteria:

1. All open Grade III tibia fractures (plateau, shaft, pilon) requiring a second procedure following fixation, or traumatic transtibial amputations requiring delayed primary closure, skin grafting and/ or flap coverage.
2. Ages 18 - 64 years inclusive
3. Patients may have risk factors for infection including diabetes, immunosuppression from steroids or other medications, HIV, or other infections.
4. Patients may have a traumatic brain injury.
5. Patients may have other fractures including spine, upper extremity fractures, contralateral lower extremity injuries, ipsilateral pelvis, hip, femur or foot injuries.
6. Patients may be treated initially at an outside institution prior to transfer to the study institution, as long as the definitive fixation was not performed prior to entrance into the study.
7. Patients with bilateral injuries that meet inclusion criteria may be included, but only the limb rated as "more severe" by the treating surgeon will be enrolled in the study.
8. Patients may have co-existing non-tibial infection, with or without antibiotic treatment.
9. Patients may have an existing infection of the surgical wound under treatment at the time of wound closure.
10. Patients may be definitively fixed using any method (nail, plate, ex fix)
11. Patients may have a fasciotomy

Exclusion Criteria:

1. Patient speaks neither English nor Spanish
2. Patient is a prisoner
3. Patient has been diagnosed with a severe psychiatric condition
4. Patient is intellectually challenged without adequate family support
5. Patient lives outside the hospital's catchment area
6. Patients with planned follow-up at another medical center

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Particiapting METRC Trauma Centers across the country.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-09 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Infection | 1 year
  The presence of a deep surgical site infection will be defined by the criteria of the Centers for Disease Control. Deep SSI occurs within 30 days after the operation if no implant is left in place, or within one year if implant is in place and the infection appears to be related to the operation.

SECONDARY OUTCOMES:
Classification of Appropriate Antibiotic Care | 1 year
  An expert panel consisting of the study PI, two additional orthopaedic trauma surgeons and at least three infectious disease experts will be convened to develop a classification grid for the most common and/or expected microbial species to be found in this study and the related antibiotic treatment regimens used in the initial care of these patients. For each microbial species, the expert panel will classify a given antibiotic regimen as "appropriate" and "not appropriate", based on the best available published data.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bosse, MD, Principal Investigator — Carolinas Medical Center
Locations (40):
- United States (40):
  - Naval Medical Center San Diego, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - University of Miami Ryder Trauma Center, Miami, Florida
  - Florida Orthopaedic Institute, Tampa, Florida
  - Emory University Dept of Orthopaedics, Atlanta, Georgia
  - OrthoIndy at St Vincent, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Louisiana State University, New Orleans, Louisiana
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Walter Reed Military Medical Center, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Orthopaedic Associates of Michigan, Spectrum Health, Grand Rapids, Michigan
  - Hennepin County Medical Center / Minneapolis, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Louis Medical Center, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Penn State University M.S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hosptial, Pittsburgh, Pennsylvania
  - Brown University/Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Miliary Medical Center, Fort Sam Houston, Texas
  - UT Health: The University of Texas Health Science Center at Houston Medical School, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Harborview Medical Center, Seattle, Washington